CLINICAL TRIAL: NCT00582270
Title: Prospective Study of Possible Infectious Disease - Associated Antigen Drive in Previously Untreated Indolent Lymphoma
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 03-012
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Indolent Non-Hodgkin's Lymphoma
Keywords: non-hodkin's lymphoma; follicular; non-follicular; infectious disease
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Follicular Lymphoma
- 2: Non-follicular Lymphoma

SUMMARY:
The purpose of this study is to determine if an infectious disease may be associated with the new lymphoma diagnosis.

Infections to be tested include:

1. Helicobacter pylori (H. pylori): This is a bacteria sometimes found in the stomach that has been associated with a particular kind of lymphoma, gastric MALT. We are interested to learn if the H. pylori infection may be associated with other indolent lymphomas.
2. Hepatitis C: This virus infection of the liver has been found in association with non-follicular lymphomas in Italy. We want to determine if the infection is associated with lymphomas in the United States.
3. Bacterial overgrowth of the small bowel: Since indolent lymphomas often affect the lymph nodes surrounding the small bowel, it may be possible that an infection within the bowel is stimulating lymphoma growth. This has never been demonstrated to date, and will be studied in this clinical study.
4. Epstein-Barr virus: This is the virus that causes infectious mononucleosis or "mono." It has been associated with other rapidly growing lymphomas, but not indolent lymphoma.

DETAILED DESCRIPTION:
This is a prospective observational clinical study of possible infectious disease-associated antigen drive in previously untreated patients with indolent lymphoma (follicular and nonfollicular cohorts).

Eligible patients with a new diagnosis of indolent lymphoma will be enrolled after informed consent. All patients will be tested for possible known infectious diseases that may contribute to antigen drive (H. Pylori; Hepatitis C), as well as for other infectious diseases not yet established as contributing to antigen drive (Borrelia; Chlamydia; and small bowel overgrowth). All patients will have a complete history recorded regarding other possible chronic infections, and an infectious disease consultation, as indicated.

Patients with positive antigen-drive infectious disease studies will be treated as indicated with standard antibiotic regimens and response (both infectious disease as well as lymphoma status)will be documented and recorded.

The primary objective of this study is (1) to evaluate the possible association of infectious diseases in previously untreated patients with indolent lymphoma. The secondary objective of this study is to evaluate possible lymphoma response the in patients treated for positive infectious disease studies; and to evaluate EBV immune responses in these previously untreated patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of follicular lymphoma: grades I, II, or IIIA, or non-follicular lymphoma: lymphoplasmacytoid lymphoma, small lymphocytic lymphoma, marginal B-cell lymphoma, or MALT lymphoma (as defined in the WHO classification2) as reviewed by a hematopathologist at Memorial Hospital.
* Staging fulfills criteria for no initial treatment according to GELF criteria for advanced stage disease. None of the following should be present: 1) a nodal or extranodal mass with a diameter of >7 cm, 2) involvement of at least three nodal sites [each with a diameter of >3 cm], 3) systemic symptoms, 4) plenomegaly, or 5) ureteral compression.
* No prior treatment for lymphoma is permitted.
* Karnofsky performance status > 70%
* The patient may not have a previous history of radiation therapy.
* Patient or guardian must be able to sign voluntary written consent.
* Male or female patients 18 years of age or greater.

Exclusion Criteria:

* Histologic diagnosis of intermediate grade or high grade non-Hodgkin's lymphoma.
* Histologic evidence of low grade transformation.
* Prior treatment for non-Hodgkin's lymphoma.
* Regional lymphoma (peripheral stages I and II) eligible for involved field irradiation.
* GELF criteria35 for institution of systemic chemotherapy, which includes: 1) a nodal or extranodal mass with a diameter of >7 cm, 2) involvement of at least three nodal sites [each with a diameter of >3 cm], 3) systemic symptoms, 4) splenomegaly, or 5) ureteral compression.
* Prior history of malignancy within the past five years or a concurrent malignancy, with the exceptions of cutaneous basal cell carcinoma or carcinoma in situ of the uterine cervix.
* Karnofsky Performance Status <70%.
* Patients with a known history of HIV seropositivity.
* Patients who require therapy with systemic corticosteroids.
* Patient or responsible guardian is unable to provide written informed consent.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Follicular and non-follicular non-Hodgkin's lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2003-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Disease status | 5 years 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Carol Portlock, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org